CLINICAL TRIAL: NCT02110589
Title: Investigation Into the Efficacy and Application of Non-invasive Sensor Technology to Produce a Community-based Seizure Alarm/Monitor for Epilepsy and Episodic Hyperexcitability Disorders.
Brief Title: Tonicity Monitor For Epilepsy and Hypertonic Disorders
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Vikel Ltd (Industry)
Collaborators: Abertawe Bro Morgannwg University NHS Trust (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: VIKEL CT001
Record Dates: First submitted 2014-04-07; First posted 2014-04-10 (Estimated); Last update posted 2014-04-10 (Estimated); Status verified 2014-04

CONDITIONS: Epilepsy
Keywords: seizures
MeSH Terms: conditions — Epilepsy; Seizures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Patient Group 1 (Experimental): Testing of Epidetect:
  Adult Patients with difficult to control tonic-clonic (convulsant) epilepsy undergoing hospitalised video telemetry monitoring. Patients will be hospitalised as part of their normal investigation of the epilepsy and patients will be consented 1 week before hospitalisation. Epidetect will be used in conjunction with the normal EEG monotoring and video telemetry. The patient will be fitted with the topical sensors at the start of monotoring and then depending on the seizure activity will wear the sensors until enough data is gathered. Hospitalisation under these circumstances typically lasts no more than five days, so monitoring with the topical sensor will be no longer than this.
  Interventions: Device: Epidetect
- Patient Group 2 (Experimental): Testing of Epidetect:
  Paediatric patients (over 7 years) where parental consent will enable the epilepsy monitor to be used at home for 1 week and brought back in for analysis along with video evidence. This will not constitute any change in normal care or treatments, and the video evidence provided represents enhanced care through accurate seizure diary reporting. Suitable families and children will be selected and consented through scheduled clinics in paediatric neurology.
  Interventions: Device: Epidetect
- Patient group 3 (Experimental): Testing of Epidetect:
  Patients where the epilepsy is suspected to be psychogenic (pseudo-seizures) rather than organic epilepsy. We will test whether the epilepsy monitor will be able to differentiate between epilepsy and psychogenic seizures in the medical setting when patients are hospitlised for seizure investigation. Suitable patients will be selected and consented through scheduled clinics in paediatric neurology (under 16) and adult neurology.
  Interventions: Device: Epidetect
- Patient Group 4 (Experimental): Testing of Epidetect:
  Internal negative Controls. Juveniles or adults with other forms of epilepsy that do not have a hypertonic (increased muscle stiffening) phenotype e.g. absence seizures.
  Interventions: Device: Epidetect
- Control Group 1 (Other): Testing of Epidetect:
  Volunteers who do not have a history of seizures / epielsy, head trauma, migraine, neurological or muscular-skeletal disorders. This is to produce the baseline data for the Monitor.
  Interventions: Device: Epidetect

INTERVENTIONS:
Device: Epidetect — Topically aplied muscle tonicity monitor (EMG recording)

SUMMARY:
Epilepsy is an episodic disorder which can result in recurrent seizures often associated with hypertonia (muscle stiffening) and myoclonia (involuntary muscle jerking). Hypertonia can often occur before full expression of the seizure and so detection of hypertonia could act as an alarm to epilepsy patients and carers in order to prepare for a seizure event. Secondly, a recording device for seizure frequency and duration is a valuable clinical tool for collecting data for clinicians who manage the disorder in primary and tertiary care. The investigators have developed a portable prototype for hypertonia detection using a non-invasive, muscle activated, sensor that records seizure activity. The investigators now want to test this sensor system in patients identified by Consultant Clinician Custodians within the Wales Epilepsy Research Network (WERN). The Epidetect® prototype has been developed by VIKEL LTD™ in collaboration with WERN - a Welsh Assembly funded network.

ELIGIBILITY:
Inclusion Criteria:

For phase 1 of the trial; - admission to the neurophysiology department at Morriston hospital for in patient video telemetry

For Phase 2 of the trial:

1. For PG-1 and PG-2 the persistence of intractable tonic-clonic epilepsy
2. For PG-3 the clinical suspicion of dissociative seizures
3. For PG-4 the clinical diagnosis of absence epilepsy
4. For CG-1 the absence of neurological, muscular-skeletal disorders
5. Suitable circumstances for informed consent in all instances

Exclusion Criteria:

For Phase 1 of the trial:

- a diagnosis of a movement disorder

For Phase 2 of the trial

1. Where learning difficulties in adult patients or carers prevents informed consent or proper home supervision in PG-2.
2. Where neurological diagnosis is ambiguous or incomplete.
3. Where topical application of the sensors causes discomfort or psychological distress.

Ages: 7 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2014-08; Primary Completion 2017-01 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Measurable changes in muscle tonicity specific to and discernable seizure activity | 2 years
  The primary outcome measure for the study will the development of a tonicity monitor that can successfully detect increases in muscle tonicity preceding a seizure event and alert the patient of an impending attack.

SECONDARY OUTCOMES:
Using the device to reliably measure seizure frequency | 2 years
Using the device to reliably measure seizure duration | 2 years
Using the device to reliably measure strength of seizure | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Inder M Sawhney, MD, FRCP, Principal Investigator — Abertawe Bro Morgannwyg University Health Board
Locations (1):
- Morriston Hospital, Swansea, United Kingdom